CLINICAL TRIAL: NCT03853382
Title: Cognitive Analytic Therapy-informed Containment for Self-Harm (CATCH): A Feasibility Trial
Brief Title: Cognitive Analytic Therapy-informed Containment for Self-Harm (CATCH)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manchester (Other)
Responsible Party: Principal Investigator, Peter Taylor, clinical lecturer, University of Manchester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 257582
Record Dates: First submitted 2019-02-20; First posted 2019-02-25 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2021-01

CONDITIONS: Self Harm
MeSH Terms: conditions — Self-Injurious Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Analytic Informed Brief Therapy (Experimental)
  Interventions: Behavioral: Cognitive analytic informed brief therapy
- Treatment As Usual (No Intervention)

INTERVENTIONS:
Behavioral: Cognitive analytic informed brief therapy — The brief CAT-informed therapy will take place over two sessions. Session one will last around 90 minutes. In session one, we will discuss with the participant their experience of self-harm and begin to support them to make sense of patterns in their self-harming behaviour. This will be done by thinking about the events that come before or follow self-harm, as well as thoughts and emotions associated with self-harm; it will also be done by thinking about ways that the participant relates to him/herself and other people. By the end of the first session, the researcher and the participant will have collaboratively developed a written diagram which shows patterns in the participant's self-harm.
  Session two will involve revisiting the mapping of patterns. The researcher and participant will the collaboratively develop 'exits' or ways to break patterns and cycles of thinking, feeling and behaviour. Both sessions will have structured endings.
  Arms: Cognitive Analytic Informed Brief Therapy

SUMMARY:
Non-suicidal self-injury (NSSI) is when somebody engages in self-harm, such as cutting, without meaning to end his or her life. A large number of people engage in NSSI for lots of reasons, for example to cope with emotions. However, currently there are large waiting lists to access psychological therapy through the NHS. Therefore, it is important to research brief therapies so that individuals who engage in NSSI can receive treatment quicker. One potentially helpful therapy suggested is Cognitive Analytic Therapy (CAT), which focuses on patterns in relationships. NSSI can be understood as a way in which people relate to themselves, which suggests that CAT would fit well in terms of understanding and working with these difficulties.

This study aims to evaluate a brief two-session CAT therapy for people who engage in NSSI. The project aims to evaluate the feasibility and acceptability of the therapy, using interviews and questionnaires. This means looking at whether participants stick with the therapy, and how they find taking part in the therapy.

All participants will meet with a researcher for an initial session to complete baseline questionnaires about their current difficulties, thoughts and feelings. Participants will then be randomly allocated to a condition: either the therapy condition or the treatment-as-usual (TAU) condition. Participants in the therapy condition will receive two therapy sessions, whilst participants in the TAU condition will not receive any therapy sessions. All participants will attend a final session to complete more questionnaires. Participants will be asked to complete online surveys weekly. Some participants will be invited to take part in interviews about their experience of the therapy. All participants will receive a shopping voucher as compensation for their time. Using the data collected from this study, future work can be done to provide better treatment for people who engage in NSSI.

ELIGIBILITY:
Inclusion Criteria:

1. Be aged over 16 years (parental consent is not needed; The British Psychological Society, 2008)
2. Be comfortable with and have access to email and the internet for completing study measures
3. Be currently under or receiving support form clinical/health service including NHS, 3rd sector, or University health services
4. Following DSM-V (American Psychiatric Association, 2013), have had five or more instances of NSSI in the past year:

   • NSSI methods are operationalised to include cutting, burning, biting, or scratching oneself, as well as head-banging or self-poisoning.
5. Have an adequate English language ability to understand study materials
6. Be deemed capable of providing informed consent by their clinical team.

Exclusion Criteria:

1. Be currently receiving any other psychological therapy (e.g. including but not limited to CBT and/or DBT), and will not have received psychological therapies in the last one month.
2. Have previously received any CAT
3. Have been diagnosed with Learning Disability or Autistic Spectrum Disorder as judged by clinical team - since the intervention has not been developed for this population
4. Be currently judged at high risk of suicidal behaviour (although if participants were keen to be involved, they could be considered when their mental health has improved).
5. Have been hospitalised as a result of self-harm in the past month

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Acceptability- attendance rates | Five weeks
  We will judge the intervention feasible based on whether > 70% of those randomised to receive the intervention complete both sessions.
Safety- adverse experiences | Five weeks
  Safety will be assessed via an Adverse Effects in Psychotherapy (AEP) self-report measure (Hutton, Byrne & Morrison, 2017; unpublished). Items rated as greater than "a little" will be classified as notable adverse experiences. Adverse events occurring during the course of the trial (identified through discussion with the participant or clinical team) will also be monitored and recorded. These will include hospitalisation (related to mental health), medically serious self-harm (i.e. requiring medical intervention), and suicidal ideation where a plan and intent are present.
Feasibility - completion rate of assessments | Five weeks
  Feasibility will be based upon (i) > 70% of participants attending the post-therapy follow-up point and (ii) a rate of missing data per outcome measure of < 25% (this rate of missing data has been used to indicate high risk of bias within systematic reviews; Hutton et al., 2015).

SECONDARY OUTCOMES:
Non-Suicidal Self-Injury | Five weeks
  Self-Injurious Thoughts and Behaviours Inventory Short-Form structured interview (SITBI-SF; Nock et al., 2007).
Self-Compassion Scale (SCS; Neff, 2003). | Five weeks
  The Self-Compassion Scale (SCS; Neff, 2003), assesses levels of self-compassion. The SCS includes 26 items rated on a scale of 1 (almost never) to 5 (almost always) as to how often participants engage in a range of thoughts or behaviours. The SCS includes six subscales including self-criticism (scores range from 5 to 25), self-kindness (scores range from 5 to 25), isolation (scores range from 4 to 20), common humanity (scores range from 4 to 20), over-identification (scores range from 4 to 20) and mindfulness (scores range from 4 to 20). Higher scores indicate greater self-compassion.
Depressive symptoms | Five weeks
  Patient Health Questionnaire (PHQ9; Kroenke et al., 2001).The PHQ9, used to assess depression, includes nine items and determines the extent to which participants have been bothered by difficulties over the last two weeks by rating on a scale of 0 (not at all) to 3 (nearly every day). Scores range from 0 to 27, with higher scores indicating greater symptom severity.
Self-concept instability | Five weeks
  The Personality Structure Questionnaire (PSQ; Pollock et al., 2001) will be used to assess self-concept stability. The PSQ includes 8 items rated on a five-point scale with opposite ends representing agreement with an unstable or stable sense of self. Scores range from 0 to 40 with greater scores indicating greater instability
Self-injury urges | Five weeks
  Alexian Brothers Urges to Self-injure scale (ABUSI; Washburn et al., 2010). The ABUSI asks participants to rate their urges to self-injure over the last week on frequency, strength, time thinking of self-injuring, and ability to resist. Score range from 0 to 30 with higher scores indicating more severe urges to self-injure

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Mersery Care NHS Foundation Trust, Liverpool
  - Greater Manchester Mental Health NHS Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: No
Due to the small scale nature of the trial there is no plan to share Individual Patient Data

REFERENCES:
- [Derived] Witt KG, Hetrick SE, Rajaram G, Hazell P, Taylor Salisbury TL, Townsend E, Hawton K. Psychosocial interventions for self-harm in adults. Cochrane Database Syst Rev. 2021 Apr 22;4(4):CD013668. doi: 10.1002/14651858.CD013668.pub2. PMID 33884617